CLINICAL TRIAL: NCT00535652
Title: Konzentrationen Von Ertapenem in Kolorektalem Gewebe
Brief Title: Concentration of Ertapenem in Colorectal Tissue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, M. Wittau, MD, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-07
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diverticulosis, Colonic; Rectal Neoplasms; Colonic Neoplasms
MeSH Terms: conditions — Diverticulosis, Colonic; Rectal Neoplasms; Colonic Neoplasms | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ertapenem (Experimental): Administration of 1 gram ertapenem I.V.
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — powder for infusion, 1 gram I.V., single dose over 30 min.
  Other Names: Invanz, EU/1/02/216/001 + /002; ATC code: J01DH03

SUMMARY:
The purpose of this study is to determine the tissue kinetics of ertapenem in colonic tissue from three hours up to six hours (25% of dosing interval) after administration of ertapenem.

DETAILED DESCRIPTION:
The purpose of this study is to determine the tissue kinetics of ertapenem in colorectal tissue from three hours up to six hours (25% of dosing interval) after administration of ertapenem before an elective surgical intervention (open or laparoscopic surgery) at the colon/rectum. Subjects are patients. Hospitalized patients 18 years or older requiring elective surgical intervention (open or laparoscopic surgery) at the colon will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients 18 years or older requiring elective surgical intervention (open or laparoscopic surgery) at the colon will be eligible for this study.
* Patients with benignant disorders (e.g. colonic diverticulosis) will be preferred.

Exclusion Criteria:

* Pregnancy or lactation in women
* Emergency surgery, history of serious allergy or intolerance to β-lactam antibiotics and other carbapenems
* Systemic antimicrobial therapy with ceftazidime (internal standard of high-performance liquid chromatography / mass spectrometry) within a 7 days period prior to study entry
* Ongoing intraabdominal infections
* Terminal illness
* Chronic immunosuppressive therapy
* Severe diseases of the liver, e.g. cirrhosis of the liver with ALT or AST > 6 x upper limit of normal (ULN) and bilirubin > 3 x ULN, severe renal insufficiency with a creatinine clearance ≤30 mL/min., neutrophil count < 1000 cells/mm3, platelets < 75000 cells/mm3 and coagulation studies (INR) > 1.5 x ULN, ongoing therapy with valproin acid.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Henne-Bruns, Prof. Dr., Principal Investigator — University of Ulm, Dept. of Visceral Surgery
Locations (1):
- University of Ulm, Dept. of Visceral Surgery, Ulm, Germany

REFERENCES:
- [Derived] Wittau M, Scheele J, Bulitta JB, Mayer B, Kaever V, Burhenne H, Henne-Bruns D, Isenmann R, Brockschmidt C. Pharmacokinetics of ertapenem in colorectal tissue. Chemotherapy. 2011;57(5):437-48. doi: 10.1159/000333377. Epub 2011 Dec 22. PMID 22189340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertapenem
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ertapenem
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 55 [25 to 76]
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 19
Region of Enrollment [Number; unit: participants]
  Germany | 23

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Ertapenem in Colorectal Tissue in mg/kg 3 to 6 Hours After a Single Dose of 1 Gram Ertapenem I.V..
Time Frame: 3 to 6 hours after a single dose of 1 gram ertapenem I.V..
Reporting Status: Not Posted

2. Secondary Outcome: Safety Assessment
Time Frame: 0 to approx. 14 days after admission
Reporting Status: Not Posted

3. Primary Outcome: Tissue (Total) Concentrations of Ertapenem in the Colorectal Tissue
Description: The mean (+- SD) tissuetotal concentrations of ertapenem in the colorectal tissue every 30 minutes up to 10 hours
Time Frame: The mean (+- SD) tissuetotal concentrations of ertapenem in the colorectal tissue as an average of every 30 miuntes up to 10 hours
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Ertapenem
Number analyzed (Participants) | 20
mg/kg | 6.4 (2.3)

ADVERSE EVENTS:
Arm/Group | Ertapenem
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ertapenem (N=20)
Urinary tract infection (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No